CLINICAL TRIAL: NCT02934269
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CC-90006 in Healthy Subjects
Brief Title: A Study of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CC-90006 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-90006-CP-001
Record Dates: First submitted 2016-10-13; First posted 2016-10-14 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
Keywords: Healthy subjects; Safety; CC-90006; Phase 1; Tolerability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- CC-90006; Dose Level 1 (Experimental): CC-90006 will be administered by subcutaneous injection in the abdomen
  Interventions: Drug: CC-90006
- CC-90006; Dose Level 2 (Experimental): CC-90006 will be administered by subcutaneous injection in the abdomen
  Interventions: Drug: CC-90006
- CC-90006; Dose Level 3 (Experimental): CC-90006 will be administered by subcutaneous injection in the abdomen
  Interventions: Drug: CC-90006
- CC-90006; Dose Level 4 (Experimental): CC-90006 will be administered by subcutaneous injection in the abdomen
  Interventions: Drug: CC-90006
- CC-90006; Dose Level 5 (Experimental): CC-90006 will be administered by subcutaneous injection in the abdomen
  Interventions: Drug: CC-90006
- Placebo (Experimental): Placebo will be administered by subcutaneous injection in the abdomen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: CC-90006
  Arms: CC-90006; Dose Level 1; CC-90006; Dose Level 2; CC-90006; Dose Level 3; CC-90006; Dose Level 4; CC-90006; Dose Level 5

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of CC-90006 following administration of single subcutaneous doses in healthy subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetic profile of single-ascending doses of CC-90006 in healthy subjects.

This will be a placebo-controlled, single-ascending dose study of CC-90006. Approximately 40 subjects will be enrolled. Five dose levels are planned. Each dose level will enroll 8 subjects who will be assigned randomly to receive active CC-90006 (6 subjects) and placebo (2 subjects).

Eligible subjects will check into the clinic site on the day before dosing (Day -1) and receive the assigned dose by subcutaneous injection the following day (Day 1). Subjects will be discharged from the site on Day 4 and return for visits on Days 8 (week 1), 15 (week 2), 22 (week 3), 29 (week 4), 36 (week 5), 43 (week 6), 57 (week 8), and 71 (week 10). Subjects will also be followed up via a phone call on Day 105 (week 15). Safety assessments will be performed and blood samples will be collected for determination of levels of CC-90006 in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, and a body mass index (BMI) of ≥ 18 and ≤ 33 kg/m2 with body weight ≥ 50 and ≤ 90 kg at screening.
* Females must have been surgically sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingo-oophorectomy; proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a follicle-stimulating hormone [FSH] level of > 40 IU/L at screening).

Exclusion Criteria:

* Exposure/treatment to an investigational (new chemical entity) or marketed drug or biologic within 30 days preceding the first dose administration, or five half-lives of that investigational drug or biologic, if known (whichever is longer).
* Donation blood or serum within 8 weeks before the first dose administration to a blood bank or blood donation center.
* History of alcohol or drug abuse (as defined by the current version of the DSM) within 2 years before the first dose administration, or positive alcohol or drug screen.
* Vaccination within 30 days prior to the first dose administration or has plans to receive a vaccination during the course of the study (including the follow phone call on Day 105).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to day 105
  Number of participants with adverse events

SECONDARY OUTCOMES:
Pharmacokinetics- Cmax | Up to day 71
  Observed maximum serum concentration
Pharmacokinetics- Tmax | Up to day 71
  Time to Observed maximum serum concentration
Pharmacokinetics- AUC0-∞ | Up to day 71
  Area under the serum concentration-time curve calculated from time zero to infinity
Pharmacokinetics- AUC0-t | Up to day 71
  Area under the serum concentration-time curve calculated from time zero to the last measured time point
Pharmacokinetics- T1/2 | Up to day 71
  Terminal half-life (T1/2)
Pharmacokinetics- CL/F | Up to day 71
  Apparent clearance of drug from serum when dosed subcutaneously
Pharmacokinetics- Vz/F | Up to day 71
  Apparent volume of distribution when dosed subcutaneously during the terminal phase
Pharmacokinetics- Anti-drug antibody | Up to day 71
  A measure of the body's immune response to CC-90006

CONTACTS AND LOCATIONS:
Overall Officials: Leon Carayannopoulos, MD, Study Director — Celgene Corporation
Locations (1):
- PPD Phase 1 Unit, Austin, Texas, United States